CLINICAL TRIAL: NCT05174039
Title: An Open-label Safety, Pharmacokinetic, and Efficacy Study of the Combination of Miglustat for the Treatment of CLN3 Disease in Patients 17 Years of Age and Older
Brief Title: An Open-label Safety, Pharmacokinetic, and Efficacy Study of Miglustat for the Treatment of Subjects With Batten Ceroid Lipofuscinosis, Neuronal 3 (CLN3) Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beyond Batten Disease Foundation (Other)
Collaborators: Theranexus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Batten-1-01
Record Dates: First submitted 2021-11-18; First posted 2021-12-30 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Batten Disease
Keywords: Batten disease; CLN3; treatment; miglustat; safety
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral miglustat (Experimental): The proposed dosing regimen is daily oral miglustat (MTD, up to 200 mg TID)
  Interventions: Drug: Miglustat 100 milligrams (mg) Oral Capsule

INTERVENTIONS:
Drug: Miglustat 100 milligrams (mg) Oral Capsule — Subjects will initiate miglustat at Week 1 and dosing will be escalated until 600mg/d. If a subject has not reached the maximum dose (600 mg/d) by Week 8, the Week 8 dose will be subject's MTD.

SUMMARY:
This is an open label study in approximately 6 subjects in 2 centers to assess the safety, PK, and efficacy of the maximum tolerable dose (MTD) of oral miglustat (100 mg once daily [QD] to 200 mg 3 times daily [TID]) in subjects ≥ 17 years of age with CLN3 disease over a period of 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

Individuals

1. Have provided informed consents (TCH and NIH) by subject or parent/legal guardian/legally authorized representative (as appropriate).
2. Are males or females ≥ 17 years of age at the time of screening
3. Have genetically confirmed diagnosis of syndromic CLN3 disease with

   EITHER:

   A. Two pathogenic mutations in the CLN3 gene, OR B. One confirmed pathogenic AND one variant of unknown significance, OR 2 variants of unknown significance, PLUS (+) secondary confirmation with evidence of characteristic inclusions on electron microscopy AND characteristic clinical course. There is no restriction on the specific CLN3 mutations for eligibility to enroll in the study. The mutations will be recorded in the electronic case report form (eCRF) for potential use in determining if CLN3 genotype is associated with tolerability and/or effectiveness of Beyond Batten Disease Foundation-1 (BBDF-1) (miglustat) therapy.
4. Male and female participants must use a highly effective method of contraception and must continue for the duration of the trial (and for 30 days after the end of treatment).
5. Are able to complete study assessments (subject or caregiver) and return to the clinic as scheduled

Exclusion criteria

Individuals

1. Have a medical condition that in the opinion of the PI would interfere with the safety assessments or increase the subject's risk of adverse events (AEs)
2. Use of any therapy (approved, off-label, or unapproved) intended to modify the course of any neuronal ceroid lipofuscinosis disease, including but not limited to flupirtine or flupirtine derivatives, cerliponase alfa (Brineura)
3. Have, in the opinion of the PI, a clinically significant abnormality in their clinical laboratory values (hematology, chemistry, or urinalysis) at screening that would preclude their participation in the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary D. Clark, MD, Principal Investigator — Texas Children Hospital; An N. Dang Do, MD, PhD, Principal Investigator — National Institute of Health Clinical Center
Locations (1):
- Texas Children Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://beyondbatten.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at hospital. The first participant was recruited on 10 March 2022 and the last participant was recruited on 08 September 2022.
Pre-assignment Details: Participants had their first enrolment visit to determine their eligibility, then a second visit within the next 42 days to confirm eligibility and perform baseline efficacy assessments. If eligibility was confirmed at the second visit, they started treatment within the next 15 days after this visit.
Groups:
- Oral Miglustat: The proposed dosing regimen was daily oral miglustat (MTD, up to 200 mg TID)
  Miglustat 100 mg Oral Capsule: participants initiated miglustat at Week 1 and dosing was to be escalated until 600mg/d. If a participant had not reached the maximum dose (600 mg/d) by Week 8, the Week 8 dose was to be participant's MTD.
Period: Overall Study
Arm/Group | Oral Miglustat
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 6
Groups:
- Oral Miglustat: The proposed dosing regimen is daily oral miglustat (MTD, up to 200 mg TID)
  Miglustat 100Mg Oral Capsule: Participants initiated miglustat at Week 1 and dosing was to be escalated until 600mg/d. If a participant had not reached the maximum dose (600 mg/d) by Week 8, the Week 8 dose will be participant's MTD.
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Body weight [Mean (Standard Deviation); unit: kilogram] | 70.45 (6.70)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter square] | 23.63 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events.
Description: Number of treatment-emergent adverse events (TEAEs) assessed at all visits and phone calls, with severity classified according to CTCAE v5.0
Time Frame: 78 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Oral Miglustat: The proposed dosing regimen is daily oral miglustat (MTD, up to 200 mg TID)
  Miglustat 100Mg Oral Capsule: Subjects will initiate miglustat at Week 1 and dosing will be escalated until 600mg/d. If a subject has not reached the maximum dose (600 mg/d) by Week 8, the Week 8 dose will be subject's MTD.
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Miglustat Pharmacokinetic (PK) Parameter Cmax
Description: Maximum plasma concentration Cmax
Time Frame: 8 weeks
Population: Descriptive statistical analyses were performed for miglustat plasma concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Oral Miglustat: The proposed dosing regimen is daily oral miglustat (MTD, up to 200 mg TID)
  Miglustat 100Mg Oral Capsule: Subjects initiated miglustat at Week 1 and dosing will be escalated until 600mg/d. If a subject had not reached the maximum dose (600 mg/d) by Week 8, the Week 8 dose was to be subject's MTD.
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
ng/ml | 2870 (35.2)

3. Secondary Outcome: Miglustat PK Parameter Tmax
Description: Time of Maximum concentration observed T max
Time Frame: 8 weeks
Population: 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
hour | 3.09 (44.1)

4. Secondary Outcome: Miglustat PK Parameter Area Under Curve (AUC)
Description: Area under the plasma concentration versus time curve Area Under Curve from pre-administration to 8 hours post-administration (AUC0-8hour). Blood draws were taken at the following time points: pre-miglustat dose (0), 1, 2, 2.5, 3, 4, 6, and 8 hours after 8 weeks of treatment.
Time Frame: 8 weeks
Population: 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
h*ng/ml | 19000 (40.3)

5. Secondary Outcome: Miglustat PK Parameter T1/2
Description: Miglustat elimination half life T1/2
Time Frame: 8 weeks
Population: 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
hour | 7.59 (19.0)

6. Secondary Outcome: Clinical Efficacy Based on Unified Batten Disease Rating Scale Subscores
Description: Change from baseline of the modified Unified Batten Disease Rating Scale (UBDRS) Physical Assessment subscale (score from 0 to 112), specifically developed to assess motor symptoms in subjects with Batten Ceroid Lipofuscinosis, Neuronal 3 (CLN3) disease. Higher scores indicate more severe disease.
Time Frame: 78 weeks
Population: 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
units on a scale | 1.76 (4.96)

7. Secondary Outcome: Clinical Efficacy With the Seizure Frequency
Description: Seizure frequency were to be assessed using a seizure diary
Time Frame: 78 weeks
Population: 6
Measure: Mean (Standard Deviation); unit: number of seizures / 3 months
Arm/Group | Oral Miglustat
Number analyzed (Participants) | 6
number of seizures / 3 months | 1.83 (3.13)

ADVERSE EVENTS:
Time Frame: Total treatment duration ranged between 510 days and 804 days, during which adverse events were collected until participants could switch to an expanded access program.
Description: The adverse event reporting focus on treatment emergent adverse events.
Arm/Group | Oral Miglustat
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Miglustat (N=6)
Dysphagia (Gastrointestinal disorders) | 1 (1) — An adverse event of Grade 3 dysphagia was diagnosed on 23 Jan 2023, 102 days after the initial dose of Batten-1 (miglustat) and 32 days after the most recent dose of study drug, considered not-related to study treatment.
Medical device site cellulitis (Infections and infestations) | 1 (1) — One hundred and one days after the initial dose of Batten-1 (miglustat) and 41 days after the most recent dose of study drug), the participant experienced Grade 3 cellulitis around the gastrostomy, leading to hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Miglustat (N=6)
Diarrhea (Gastrointestinal disorders) | 6 (19)
Weight decreased (Investigations) | 6 (17)
Tremor (Nervous system disorders) | 5 (9)
Influenza-like illness (General disorders) | 5 (6)
Seizure (Nervous system disorders) | 4 (78)
Anxiety (Psychiatric disorders) | 4 (4)
Platelet count decreased (Investigations) | 3 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (5)
Flatulence (Gastrointestinal disorders) | 3 (4)
Anal incontinence (Gastrointestinal disorders) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Lethargy (Nervous system disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (5)
Urinary incontinence (Renal and urinary disorders) | 2 (4)
Drooling (Nervous system disorders) | 2 (3)
Myoclonus (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized tonic-clonic seizures (Nervous system disorders) | 1 (4)
Nervous system disorder (Nervous system disorders) | 1 (4)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Blood creatinine phosphokinase increased (Investigations) | 1 (2)
Dysarthria (Nervous system disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrage (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Weight increase (Investigations) | 1 (1)
Electrocardiogram P Wave abnormal (Investigations) | 1 (1)
Vitamine B12 increased (Investigations) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Loss of proprioception (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Infected bite (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung opacity (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypoacousis (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT05174039/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05174039/SAP_001.pdf